CLINICAL TRIAL: NCT01105338
Title: Lycopene or Green Tea a Feasibility Study in Men at Risk of Prostate Cancer
Brief Title: Lycopene or Green Tea for Men at Risk of Prostate Cancer
Acronym: ProDiet
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Bristol (Other)
Responsible Party: Principal Investigator, Dr Athene Lane, Study Coordinator and Senior Research Fellow, University of Bristol
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C11046/A10052; ISRCTN-95931417 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tea; Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Green tea drink (Active Comparator): Green tea drink
  Interventions: Behavioral: Green tea drink
- Green tea capsules (Active Comparator): Green tea capsules
  Interventions: Dietary Supplement: green tea capsules
- Green tea placebo capsules (Placebo Comparator): Green tea placebo capsules
  Interventions: Other: Green tea placebo capsules
- Lycopene capsules (Active Comparator): Lycopene capsules
  Interventions: Dietary Supplement: Lycopene capsules
- Lycopene placebo capsules (Placebo Comparator): Lycopene placebo capsules
  Interventions: Other: Lycopene placebo capsules
- Tomato rich diet (Active Comparator): Tomato rich diet
  Interventions: Other: Tomato rich diet

INTERVENTIONS:
Behavioral: Green tea drink — Green tea drink
  Arms: Green tea drink
Dietary Supplement: green tea capsules — green tea capsules
  Arms: Green tea capsules
Other: Green tea placebo capsules — Green tea placebo capsules
  Arms: Green tea placebo capsules
Dietary Supplement: Lycopene capsules — Lycopene capsules
  Arms: Lycopene capsules
Other: Lycopene placebo capsules — Lycopene placebo capsules
  Arms: Lycopene placebo capsules
Other: Tomato rich diet — Tomato rich diet
  Arms: Tomato rich diet

SUMMARY:
RATIONALE: Lycopene and green tea may stop or delay the development of recurrent prostate cancer in patients has been treated for prostate cancer. It is not yet known whether lycopene or green tea may be more effective in preventing prostate cancer.

PURPOSE: This randomized phase II trial is studying lycopene to see how well it works compared with green tea in preventing prostate cancer in patients previously enrolled in the ProtecT trial

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess serum lycopene and epigallocatechin-3-gallate (green tea) levels at 6 months following randomization in patients with prostate cancer previously enrolled on ProtecT

Secondary

* To evaluate trial recruitment and randomization rates of patients treated with this regimen.
* To evaluate intervention tolerability in patients treated with this regimen.
* To evaluate compliance of patients treated with this regimen.
* To evaluate trial retention of patients treated with this regimen.
* To assess PSA values in patients treated with this regimen.
* To evaluate dietary compliance with recommendations of patients treated with this regimen.
* To assess weight and body mass index of patients treated with this regimen.
* To evaluate attitudes and views of men and their spouses about dietary modification and participation in long-term study.

OUTLINE: Patients are stratified according to PSA test levels obtained from ProtecT study recruitment clinic (< 3.0 ng/mL vs 3.0-19.99 ng/mL). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
Inclusion criteria: PSA level 2.0-2.95 ng/mL OR PSA level ≥ 3.0 ng/mL with a negative biopsy No major comorbidities No other cancers or prior prostate malignancy No history of allergic reactions to green tea or lycopene-containing products, including guava or watermelon Exclusion criteria: No concurrent finasteride or dutasteride

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Serum lycopene and epigallocatechin-3-gallate (green tea) levels at 6 months following randomization | 6 months

SECONDARY OUTCOMES:
Trial recruitment and randomization rates at each stage of the study | 6 months
Intervention tolerability (adverse event reporting during the six months of follow-up) | 6 months
Compliance (returned tablet counts and self-reported counts at 6 months) | 6 months
Trial retention (participants completing 6-month follow-up and questionnaires) | 6 months
PSA values at baseline and at 6 months | 6 months
Dietary compliance with recommendations (dietary questionnaire completed at 6 months and participant data reporting dietary change) | 6 months
Weight and body mass index at 1 and 6 months | 6 months
Blood pressure at 1 and 6 months | 6 months
Attitudes and views of men and their spouses about dietary modification and participation in long-term study (qualitative interviews conducted throughout the study) | 6 months
Anxiety, depression, and psychological state as measured by the Hospital Anxiety and Depression Scale and the Profile of Moods States | 6 months
Urinary symptoms as measured by the ICSmaleSF questionnaire (including voiding and incontinence scores, nocturia, frequency, and urinary-specific quality-of-life care data sources) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Athene Lane, PhD, Principal Investigator — University of Bristol
Locations (1):
- Southmead Hospital, Bristol, England, United Kingdom